CLINICAL TRIAL: NCT04593433
Title: A 3-month Cycle of Virtual Weekly Montreal Museum of Fine Arts Tours to Promote Social Inclusion, Well-being, Quality of Life and Health in Older Community Members : a Pilot Study
Brief Title: A 3-month Cycle of Virtual Guided Tours to Promote Health in Older Community Members in a Context of COVID-19 Induced Social Isolation: a Pilot Study
Acronym: VGV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal Investigator, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-2604
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Social Isolation; Quality of Life; Well Aging; Frailty
MeSH Terms: conditions — Social Isolation; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Group with the virtual museum guided tours
  Interventions: Other: Museum virtual guided tours

INTERVENTIONS:
Other: Museum virtual guided tours — The intervention is a participatory art-based activity which consists in MMFA virtual guided tours. Each virtual guided tour is performed with a group of 5 participants. They meet online one time per week for a 20 to 25 min of a visit tour during a 3-month period. Each tour is different and supervised by a MMFA trained guide.

SUMMARY:
Social isolation is defined as the objective and/or subjective reduction of number and quality of interpersonal contacts leading to a loss of an individual's social role and stigmatization. It is a major problem in Canadian society with a high prevalence in the older population (30% in individuals aged 65 and over, representing 1.5 million individuals). Social isolation is associated with a wide range of mental and physical health problems that leads to an increase in the use of health and social services. This issue increased with the coronavirus disease (COVID-19) pandemic which attacking your society at its core. Social distancing and in particular home confinement exacerbated social isolation of frailer groups like the elderly people.

In 2016, the International Federation on Ageing reported that "the main new problem facing seniors in Canada is maintaining their social contacts and activities". This highlights the need for efficient and effective interventions to improve the social inclusion of older adults experiencing social isolation.

Research suggests that art-based activities carried out at museums have significant benefits for older adults experiencing social isolation, and may foster social inclusion, well-being, quality of life and mitigate frailty. Yet few studies have examined empirically the effects of museum art-based activities in older adults experiencing social isolation. In 2019, the principal investigator of this research conducted an experimental pilot study based on a pre-post intervention (i.e., 3-month cycle of weekly guided tours carried out at the Montreal Museum of Fine Arts (MMFA)), single arm, prospective and longitudinal follow-up named "Effects of Montreal Museum of Fine Arts visits and older community dwellers with a precarious state: An experimental study", which indicated the potential of museum tours to improve social inclusion, well-being, the quality of life and frailty in older community members experiencing social isolation.

However, these studies were performed before the COVID-19 crisis and were in-site activities. The principal investigator hypothesizes that a 3-month cycle of virtual weekly MMFA tours may induce changes in well-being, quality of life and health condition in older community dwellers participating like the 'Beautiful Thursday' cycle, and that this activity can prevent the worsening of vulnerability and social isolation due to social distancing.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years and over
* Having an Internet access and an electronic device (smartphone and/or tablet) at the participant's place of living as the repetitive assessments for this study will be performed on the web platform of the Centre of Excellence on Longevity of McGill University, and the guided tours will be virtual.
* Understanding and writing the language of the recruitment centre (i.e., French or English)

Exclusion Criteria:

* a concomitant participation to an experimental study,
* planning to have a journey over one week during the cycle of visits,
* having participated to a participatory art-based activity of the MMFA during the 6 month-period before the recruitment,
* not speaking the language of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
Well-being | 3 months
  using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) self-validated questionnaire composed by 14 positively worded item scale with five response categories. It covers most aspects of positive mental health (positive thoughts and feelings). Scores can range from a minimum of 14 to a maximum of 70 points. Higher scores are associated with higher levels of mental well-being
Quality of life | 3 months
  using EuroQol-5D (EQ-5D), a standardized measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. It is composed of two parts: a questionnaire of five questions with score per question ranged from 1 (i.e., no issue) to 5 (i.e., worse issue), each question ranged from 0 (i.e., no issue) to 25 (i.e., worse issue), and a visual analogic scale of how good or bad participant health was. This scale is numbered from 0 (i.e., worse health participant can imagine) to 100 (i.e., best health participant can imagine).
frailty | 3 months
  using CESAM questionnaire, composed of 20 items providing two complementary information: 1) A global score of frailty ranged from 0 (i.e., best health and functional condition) to 18 (i.e., worse health and functional condition) and 2) Categorized health condition in four levels (vigorous with a score between 0 and 3, mild frailty with a score between 4 and 7, moderate frailty with a score between 8 and 12, and important frailty with a score above 12).
social isolation | 3 months
  using the digital form of the 11-item Dike Social Support Index (DSSI). The index is composed of two subscales: social interaction (i.e., frequency of interactions) and subjective support (i.e., satisfaction with emotional support provided). DSSI score ranges from 11 to 33, increased score indicating higher levels of social insertion. The scores of the 11 items are combined and categorized as low-fair (score ≤26), high (score 27-29) and very high (score 30-33). We will use the mean score of 11-item DSSI and its distribution in three categories.
socio-geriatric vulnerability | 3 months
  using ESOGER questionnaire, composed of 17 items exploring the COVID risk, the COVID past history, the social isolation risk due to COVID (access to food, home support and healthcare, contact with external persons, anxiety). Items correspond to a question in closed-ended format (i.e., yes or no, or calling for a specific answer). The ESOGER categorizes state of vulnerability in three levels (Low, Moderate and High vulnerability).

SECONDARY OUTCOMES:
Incident planned and unplanned visits to physicians, Emergency Department (ED) and hospitalization | 3 months
  recorded at the end of the cycle by asking directly to the participants
compliance | 3 months
  determined by the total number of guided tours performed, on a maximum of 12.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada